CLINICAL TRIAL: NCT00582829
Title: Colorectal Cancer Screening Intervention for Family Members of Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fox Chase Cancer Center (Other); Icahn School of Medicine at Mount Sinai (Other); Lombardi Comprehensive Cancer Center (Other); Micromass Communications, Cary, NC (Unknown); University of Pennsylvania (Other); Christiana Care Health Services (Other); Pinnacle Health Regional Cancer Center, Harrisburg, PA (Unknown); Temple University (Other); St. Mary Regional Cancer Center, Langhorne, PA (Unknown); South Jersey Regional Cancer Center, Bridgton, New Jersey (Unknown); Hunterdon Cancer Center (Unknown); Northeast Regional Cancer Institute (Other); Virtua Memorial Hospital and Virtua West (Unknown); Jersey Hospital (Unknown); Rutgers Cancer Institute of New Jersey (Other); Massachusetts General Hospital (Other); Main Line Health (Other); Roswell Park Cancer Institute (Other); HematologyOncology (Unknown); Associates of Central New York (Unknown); Augusta University (Other)
Responsible Party: Arnold Markowitz, Memorial Sloan Kettering Cancer Center
Other Study IDs: 03-043
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal; Cancer; Screening; Intervention
Keywords: Colorectal; Cancer; Screening; Intervention; Family
MeSH Terms: conditions — Neoplasms

GROUPS / COHORTS (3):
- 1: Generic Print Intervention: The generic print intervention will consist of the pamphlet, "Colorectal Cancer Screening Saves Lives" published by the Center for Disease Control that will be mailed to the participant.
  Interventions: Other: Generic Print Intervention
- 2: Tailored Print Intervention: The tailored print intervention will consist of a cover letter detailing the participant's stage of readiness along with a color pamphlet with information personally tailored for the individual participant.
  Interventions: Other: Tailored Print Intervention
- 3: Tailored print plus tailored phone intervention: The tailored print plus tailored telephone intervention will consist of a phone counseling session and the tailored print information described above. The tailored print material will serve as a guide during the telephone counseling contact and a reinforcement of the information.
  Interventions: Other: Tailored print plus tailored phone intervention

INTERVENTIONS:
Other: Generic Print Intervention — Generic Print Intervention: The generic print intervention will consist of the pamphlet, "Colorectal Cancer Screening Saves Lives" published by the Center for Disease Control that will be mailed to the participant.
  Groups: 1
Other: Tailored Print Intervention — Tailored Print Intervention: The tailored print intervention will consist of a cover letter detailing the participant's stage of readiness along with a color pamphlet with information personally tailored for the individual participant.
  Groups: 2
Other: Tailored print plus tailored phone intervention — Tailored print plus tailored phone intervention: The tailored print plus tailored telephone intervention will consist of a phone counseling session and the tailored print information described above. The tailored print material will serve as a guide during the telephone counseling contact and a reinforcement of the information.
  Groups: 3

SUMMARY:
This proposed study will use previous study results to guide the development and evaluation of interventions to improve CRC screening acceptance. The proposed study will evaluate the impact of three interventions to promote CRC screening among siblings in this increased-risk group, who are not currently compliant with CRC screening guidelines: 1) a generic print intervention; 2) a tailored print intervention, and; 3) a tailored print plus tailored telephone counseling intervention.

DETAILED DESCRIPTION:
First-degree relatives of individuals with CRC are at increased-risk of developing colorectal cancer (CRC). For these increased-risk individuals current guidelines recommend initiating CRC screening a decade earlier than for those at average-risk for CRC; thus, starting at age 40, or 10 years younger than the age at which the affected relative was diagnosed with CRC. In our prior study of 504 at-risk siblings of patients with a history of CRC, diagnosed at age less than 56, we found that approximately 44% of these siblings were not compliant with CRC screening guidelines. Guided by the Transtheoretical, Health Belief and Dual Process models, our prior study identified key attitudinal and non-attitudinal predictors of screening behaviors and intentions.

This proposed study will use these results to guide the development and evaluation of interventions to improve CRC screening acceptance. The proposed study will evaluate the impact of three interventions to promote CRC screening among siblings in this increased-risk group, who are not currently compliant with CRC screening guidelines: 1) a generic print intervention; 2) a tailored print intervention, and; 3) a tailored print plus tailored telephone counseling intervention.

Siblings in the generic print condition will receive a pamphlet about colorectal cancer screening published by the Center for Disease Control. Siblings in the tailored print and telephone counseling conditions will receive messages tailored specifically to their responses on targeted attitudinal and non-attitudinal measures. Five hundred twenty four siblings meeting eligibility criteria will be randomly assigned to one of the three conditions after a baseline interview assessing CRC screening behaviors and attitudes, and it is anticipated that 427 siblings will complete the study. For siblings in the tailored conditions, baseline information will be utilized to design the tailored messages. After receiving the intervention information, participants will be interviewed again six months later regarding CRC screening behaviors and attitudes to assess the impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* How old is the participant? (≥ 18 years)
* Is the participant either:
* currently age 40 or above (YES) OR
* within 10 years of the age at which the patient/proband was initially diagnosed with CRC (whichever is the younger age) (YES)
* Is the participant a full or half biological sibling of the patient/proband? (YES)

Exclusion Criteria:

* Is the participant currently not compliant with standard CRC screening guidelines? (NO)
* Is the participant English speaking? (YES)
* Does the participant have a primary language other than English? (NO)
* Does the participant have a history of Inflammatory Bowel Disease? (NO)
* Does the participant have a history of colorectal cancer of colorectal polyp? (NO)
* Does the participant have a history of hereditary colorectal cancer syndrome? (Familial Adenomatous Polyposis or Hereditary Nonpolyposis Colorectal Cancer) (NO)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Phone follow-up interview. Participants will be contacted by study assistant and the survey administered. | 6 months after baseling

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Markowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States